CLINICAL TRIAL: NCT01824940
Title: Sanitation, Hygiene, Infant Nutrition Efficacy Project
Brief Title: SHINE Sanitation, Hygiene, Infant Nutrition Efficacy Project
Acronym: SHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Ministry of Health and Child Welfare, Zimbabwe (Other); Zvitambo (Other); Cornell University (Other); University of London (Other); Bill and Melinda Gates Foundation (Other); Department for International Development, United Kingdom (Other Government); Wellcome Trust (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jean Humphrey, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB00004205; R01HD060338 (NIH)
Record Dates: First submitted 2012-03-27; First posted 2013-04-05 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Growth; Stunting, Nutritional; Anemia
Keywords: Cluster randomized trial; Nutrition; Water Sanitation Hygiene; Environmental enteropathy
MeSH Terms: conditions — Growth Disorders; Anemia | interventions — Standard of Care; Nutritional Status; Therapeutic Irrigation

STUDY DESIGN:
Masking Description: Given the nature of the intervention, masking to treatment group is not possible.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard of Care (Placebo Comparator): The Standard of Care interventions are the blanket interventions.
  Interventions: Behavioral: Standard care
- WASH (Active Comparator): One of two active interventions to be studied in this 2X2 (two by two) Factorial trial:
  Intervention 1: a package of interventions to improve household sanitation and hygiene (WASH)
  Interventions: Other: WASH
- Nutrition (Active Comparator): One of two active interventions to be studied in this 2X2 Factorial trial:
  Intervention 2: a package of interventions to improve infant and young child feeding (IYCF)
  Interventions: Dietary Supplement: Infant and young child feeding
- WASH and Nutrition (Active Comparator): This arm receives a combination of all standard care interventions, all WASH and all IYCF interventions.
  Interventions: Other: WASH and Nutrition

INTERVENTIONS:
Behavioral: Standard care — Standard Care:
  * Exclusive breastfeeding promotion for all infants, birth to 6 months
  * Strengthened PMTCT (prevention of mother to child transmission of HIV) services
  * Strengthened Village Health Worker system
  Arms: Standard of Care
Other: WASH — WASH:
  * Standard care interventions
  * Provide household ventilated pit latrine, water treatment solution, and monthly liquid soap, two hand-washing facilities and protected infant play space
  * Provide interpersonal communication interventions promoting feces disposal in a latrine, HWWS (hand washing with soap), drinking water treatment, hygienic weaning food preparation, and preventing babies from putting dirt and animal feces in their mouths.
  Arms: WASH
Dietary Supplement: Infant and young child feeding — IYCF:
  * Standard care interventions
  * Provide 20 g/d Nutributter from 6-18 months
  * Provide interpersonal communication interventions promoting optimal use of locally available foods for complementary feeding after 6 months, continued breastfeeding and feeding during illness.
  Other Names: Nutrition
  Arms: Nutrition
Other: WASH and Nutrition — WASH AND IYCF interventions
  * Standard care interventions
  * All WASH interventions
  * All IYCF interventions
  Other Names: WASH and IYCF
  Arms: WASH and Nutrition

SUMMARY:
Globally, stunting affects 26% (165 million) of under-5-year children, underlies 15-17% of their mortality and leads to long-term cognitive deficits, fewer years and poorer performance in school, lower adult economic productivity, and a higher risk that their own children will also be stunted, perpetuating the problem into future generations. Stunting begins antenatally and peaks at 18-24 months of postnatal life, when mean length-for-age Z-score (LAZ) is about -2.0 among children living in Africa and Asia. Improving the diets of young children can reduce stunting, though, at best, only by about one-third. Frequent diarrheal illness has also been implicated. However, the effect of diarrhea on permanent stunting is relatively small, maybe because children grow at "catch-up" rates between illness episodes.

The Sanitation Hygiene Infant Nutrition Efficacy (SHINE) trial is motivated by a 2-part premise:

* A major cause of child stunting and anemia is Environmental Enteric Dysfunction (EED). EED is a subclinical disorder of the small intestine, which is virtually ubiquitous among asymptomatic people living in low-income settings throughout the world. EED is characterized by increased permeability which facilitates microbial translocation into the systemic circulation and triggers chronic immune activation.
* The primary cause of EED is infant ingestion of fecal microbes due to living in conditions of poor quality and quantity of water, sanitation, and hygiene (WASH).

DETAILED DESCRIPTION:
The Sanitation Hygiene Infant Nutrition Efficacy ("SHINE") trial will test the effects of two packages of interventions: 1) improved water, sanitation and hygiene (WASH) and 2) improved infant and young child feeding (IYCF) on child stunting and anemia in the first 18 months of life. The trial will be conducted in rural Zimbabwe where WASH is poor, food insecurity high, and where about 15% of pregnant women are infected with HIV. The study will enroll 5282 women early in pregnancy and follow them and their infants until 18 months after delivery. The study will be a cluster-randomized controlled trial: two entire districts in central Zimbabwe have been divided into 212 geographic areas, each of about 100 households. The areas will be randomly allocated (that is, assigned by according to chance like the flip of a coin) to one of four interventions:

1. Improved WASH (a ventilated pit latrine, hand washing facilities with soap, drinking water treatment, a protected play space and health lessons to adopt improved hygiene behaviors)
2. Improved Infant Nutrition (health lessons on best infant feeding practices and a nutritional supplement (Nutributter) to be fed daily to babies from 6 to 18 months).
3. Improved WASH and Infant Nutrition (both interventions)
4. Standard of Care

All women living in the two districts who become pregnant during the recruitment period of the study will be invited to enroll. They will receive one of the 4 packages of interventions according to the area where they live. Health lessons will be given by Village Health Workers. Latrines and hand washing facilities will be constructed by building teams. Mothers will be followed up by research nurses at 7 months gestation, and at 1, 3, 6, 12, and 18 months after delivery. Primary outcomes are infant height and hemoglobin at 18 months of age.

Within SHINE we will measure two causal pathways: the biomedical pathway and the program impact pathway.

The biomedical pathway comprises the infant biologic responses to the WASH and IYCF interventions that ultimately result in attained stature and hemoglobin concentration at 18 months of age; it will be elucidated by measuring biomarkers of intestinal structure and function (inflammation, regeneration, absorption and permeability); microbial translocation; systemic inflammation; and hormonal determinants of growth and anemia among a subgroup of infants enrolled in an EED substudy. The investigators will also ask these mothers to record daily any episodes of diarrhea; blood/mucus in the stool; cough; fast or difficult breathing; fever; and lethargy preventing breastfeeding, that the child has between 1 month and 18 months of age. A subgroup of infants will also have stool samples collected during diarrhoeal episodes to evaluate reductions in pathogen-specific diarrhoea following WASH interventions.

Since the mothers enrolled in SHINE will have lived in unsanitary living conditions throughout their lives, it is anticipated that most will have some degree of EED themselves. It is hypothesized that resulting chronic inflammation contributes to adverse birth outcomes, such as prematurity and low birth weight. This question will be investigated through an observational design. For all mothers enrolled in SHINE, the sugar absorption test described above will be conducted and specimens of saliva, stool and blood collected and archived at the 10-12 week gestation visit for subsequent assessment of EED biomarkers. The association of severity of EED with risk of adverse birth outcomes (low birth length and weight; miscarriage, stillbirth, and premature delivery) will be assessed.

The program impact pathway comprises the series of processes and behaviors linking implementation of the interventions with the two child health outcomes; it will be modeled using measures of fidelity of intervention delivery and household uptake of promoted behaviors and practices. We will also measure a range of household and individual characteristics, social interactions, and maternal capabilities for childcare, which we hypothesize will explain heterogeneity along these pathways.

ELIGIBILITY:
Study participants will be women who are rural residents of Chirumanzu or Shurugwi districts in Zimbabwe and who become pregnant during the enrollment period of the trial and are identified and consent to participation during pregnancy, and their live born infants. A total of 5280 women will be enrolled.

Inclusion Criteria:

Pregnant women residing in the study districts, whose pregnancy is confirmed by a urine pregnancy test.

Exclusion Criteria:

* Women residing in the study districts who become pregnant during the enrollment period but do not consent to join the trial
* Women who reside in urban areas of these two districts
* Infants with major non-fatal abnormalities will not be excluded from study procedures, but will be excluded from the final analytic sample if the abnormality is likely to directly affect gut health/function or stature (e.g. neural tube defects, cerebral palsy, Down syndrome)

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5280 (Actual)
Dates: Start 2012-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Infant length at 18 months | 18 months of age. Protocol and Statistical Analysis Plan are available at https://osf.io/w93hy.
  Recumbent length measured by length board
Infant hemoglobin at 18 months | 18 months
  Measured by Hemocue

SECONDARY OUTCOMES:
Infant environmental enteric dysfunction | 1, 3, 6, 12 and 18 months of age
  Assessed in a subgroup of infants recruited to the EED substudy by assessing domains of the hypothesized EED pathway using biomarkers of intestinal structure and function (inflammation, regeneration, absorption and permeability); microbial translocation; systemic inflammation; and hormonal determinants of growth and anemia
Infant weight, mid-upper arm circumference and head circumference | At 18 months, and (with length) at intermediate time-points of 1, 3, 6 and 12 months
  Measured by standardized anthropometry protocols at each age
To describe the Program Impact Pathways (PIP) linking implementation of each randomized intervention (WASH and IYCF) with length and hemoglobin concentrations | Throughout follow-up
  Assessment of quality of VHW training and supervision; VHW Capacity, defined as a composite of attained knowledge, goal setting capacity, and achieved performance; Fidelity of intervention implementation, defined as degree of conformance with protocol specifications for both VHW and mother; Attained maternal knowledge and skills assessed by questionnaire and observation; Uptake or adoption of promoted behaviors by mothers and their households assessed by questionnaire and observation.
Exclusive breastfeeding | First 6 months of life
  To describe the prevalence of exclusive breastfeeding among all infants enrolled in the trial by maternal/infant HIV status.
To evaluate the effect of the IYCF intervention on uptake of improved infant feeding practices by maternal/infant HIV status | 6-18 months of age
  Infant diet quality as assessed by World Health Organization IYCF indicators ; infant nutrient intake from complementary foods assessed by 24 hour dietary recall; appropriate use of Nutributter from 6 to 18 months.
To evaluate the effect of the WASH intervention on the 5 key behaviors it promotes by maternal/infant HIV status | Throughout follow-up
  Proper disposal of animal and human feces; Handwashing with soap after fecal contact; Point-of-use chlorination of drinking water; Protecting children from ingestion of dirt and feces; Feeding baby freshly prepared foods, or reheating leftover food.
Relative contributions of diarrhea vs EED | Birth to 18 months
  To model the relative contributions of diarrheal disease and EED in mediating the effects of improved WASH on child length and hemoglobin concentrations, stratified by maternal/infant HIV status.
To measure the strength of association between other potential causes of stunting and anemia (other than poor WASH or IYCF) with linear growth and hemoglobin | Throughout follow-up
  Maternal schistosomiasis infection during pregnancy; Maternal HIV infection together with adherence to antiretroviral and cotrimoxazole regimens during pregnancy and lactation; Infant HIV infection or exposure, together with adherence to antiretroviral and/or cotrimoxazole regimens; Exposure to dietary mycotoxin contamination by the mother during pregnancy and lactation, and by the infant during complementary feeding.
Infant diarrhea prevalence, incidence and severity | 1 month to 18 months of age
  Assessed by 7-day morbidity history in all infants, and by daily morbidity diary in a subgroup of infants
Child neurodevelopment | 24 months of age
  Assessed by MacArthur-Bates Communication Developmental Inventory; Malawi Development Test (MDAT); A not B task; Delayed inhibition task; and Caregiver Child Interaction assessment in a subgroup of children
Prevalence of mycotoxin exposure among mothers and infants | Maternal samples assessed at baseline; infant samples assessed birth to 18 months
  Detectable AFB1-lysine in plasma and detectable AFM1 in urine; detectable Fumonisin B1 in urine; detectable deoxynivalenol in urine; detectable zearalenone in urine; detectable ochratoxin A in urine; detectable T-2 in urine
MAternal and infant microbiota | Maternal samples from baseline and 1 month postpartum; infant samples birth to 18 months of age
  16S rRNA and whole genome sequencing of DNA and RNA from stool to define th composition and function of the microbial community that inhabits the human intestine.
Infant rotavirus vaccine and polio vaccine immunogenicity | 1 and 3 months of age
  Measurement of rotavirus IgA titre in plasma, measurement of polio virus IgA titre in plasma
Adverse birth outcomes: miscarriage, still birth, small for gestational age, preterm delivery, neonatal death | Maternal pregnancy exposures, infant outcomes through 1 month postpartum
  Association of maternal exposures during pregnancy (EED, anemia, mycotoxin exposure, HIV infection, schistosomiasis infection) on each adverse birth outcome
Bioimpedance analysis, skinfold thicknesses and leg length measurement | 24 months in a subsample of infants
  Assess the impact of the randomized interventions on infant body composition. analysis plan at https://osf.io/t9zd4
Observational study of WASH and non-WASH infants | About 14 months of age
  90 WASH and 90 non-WASH infants will undergo 6 h structured observation to directly observe and assess intervention impact on hygiene behaviors
Assess metabolic pathways of pathogenesis of stunting | 12 month urines; longitudinal stools from 150 mother-infant pairs from 32 week gestation, and 1,3,6,12,and 18 months postpartum
  Urine and stool samples analysed by untargeted metabolomics
Friendship Bench for treatment of depression: a pilot study | August 2018 - January 2019 (about a year after the end of the trial).
  30 SHINE mothers will be recruited to pilot a depression intervention for feasibility and acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Jean H Humphrey, ScD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (1):
- Zvitambo, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Humphrey JH. Child undernutrition, tropical enteropathy, toilets, and handwashing. Lancet. 2009 Sep 19;374(9694):1032-1035. doi: 10.1016/S0140-6736(09)60950-8. No abstract available. PMID 19766883
- [Background] Prendergast AJ, Rukobo S, Chasekwa B, Mutasa K, Ntozini R, Mbuya MN, Jones A, Moulton LH, Stoltzfus RJ, Humphrey JH. Stunting is characterized by chronic inflammation in Zimbabwean infants. PLoS One. 2014 Feb 18;9(2):e86928. doi: 10.1371/journal.pone.0086928. eCollection 2014. PMID 24558364
- [Background] Paul KH, Muti M, Chasekwa B, Mbuya MN, Madzima RC, Humphrey JH, Stoltzfus RJ. Complementary feeding messages that target cultural barriers enhance both the use of lipid-based nutrient supplements and underlying feeding practices to improve infant diets in rural Zimbabwe. Matern Child Nutr. 2012 Apr;8(2):225-38. doi: 10.1111/j.1740-8709.2010.00265.x. Epub 2010 Aug 4. PMID 22405701
- [Background] Mbuya MN, Humphrey JH, Majo F, Chasekwa B, Jenkins A, Israel-Ballard K, Muti M, Paul KH, Madzima RC, Moulton LH, Stoltzfus RJ. Heat treatment of expressed breast milk is a feasible option for feeding HIV-exposed, uninfected children after 6 months of age in rural Zimbabwe. J Nutr. 2010 Aug;140(8):1481-8. doi: 10.3945/jn.110.122457. Epub 2010 Jun 23. PMID 20573941
- [Background] Ngure FM, Humphrey JH, Mbuya MN, Majo F, Mutasa K, Govha M, Mazarura E, Chasekwa B, Prendergast AJ, Curtis V, Boor KJ, Stoltzfus RJ. Formative research on hygiene behaviors and geophagy among infants and young children and implications of exposure to fecal bacteria. Am J Trop Med Hyg. 2013 Oct;89(4):709-16. doi: 10.4269/ajtmh.12-0568. Epub 2013 Sep 3. PMID 24002485
- [Background] Mupfudze TG, Stoltzfus RJ, Rukobo S, Moulton LH, Humphrey JH, Prendergast AJ; SHINE Project Team. Hepcidin decreases over the first year of life in healthy African infants. Br J Haematol. 2014 Jan;164(1):150-3. doi: 10.1111/bjh.12567. Epub 2013 Sep 20. No abstract available. PMID 24112078
- [Background] Ngure FM, Reid BM, Humphrey JH, Mbuya MN, Pelto G, Stoltzfus RJ. Water, sanitation, and hygiene (WASH), environmental enteropathy, nutrition, and early child development: making the links. Ann N Y Acad Sci. 2014 Jan;1308:118-128. doi: 10.1111/nyas.12330. PMID 24571214
- [Background] Palha De Sousa CA, Brigham T, Chasekwa B, Mbuya MN, Tielsch JM, Humphrey JH, Prendergast AJ. Dosing of praziquantel by height in sub-Saharan African adults. Am J Trop Med Hyg. 2014 Apr;90(4):634-7. doi: 10.4269/ajtmh.13-0252. Epub 2014 Mar 3. PMID 24591432
- [Background] Gough EK, Moodie EE, Prendergast AJ, Johnson SM, Humphrey JH, Stoltzfus RJ, Walker AS, Trehan I, Gibb DM, Goto R, Tahan S, de Morais MB, Manges AR. The impact of antibiotics on growth in children in low and middle income countries: systematic review and meta-analysis of randomised controlled trials. BMJ. 2014 Apr 15;348:g2267. doi: 10.1136/bmj.g2267. PMID 24735883
- [Background] Desai A, Mbuya MN, Chigumira A, Chasekwa B, Humphrey JH, Moulton LH, Pelto G, Gerema G, Stoltzfus RJ; SHINE Study Team. Traditional oral remedies and perceived breast milk insufficiency are major barriers to exclusive breastfeeding in rural Zimbabwe. J Nutr. 2014 Jul;144(7):1113-9. doi: 10.3945/jn.113.188714. Epub 2014 May 14. PMID 24828026
- [Background] Jones AD, Rukobo S, Chasekwa B, Mutasa K, Ntozini R, Mbuya MN, Stoltzfus RJ, Humphrey JH, Prendergast AJ. Acute illness is associated with suppression of the growth hormone axis in Zimbabwean infants. Am J Trop Med Hyg. 2015 Feb;92(2):463-70. doi: 10.4269/ajtmh.14-0448. Epub 2014 Dec 22. PMID 25535308
- [Background] Mupfudze TG, Stoltzfus RJ, Rukobo S, Moulton LH, Humphrey JH, Prendergast AJ; SHINE Trial Team; Jones AD, Manges A, Mangwadu G, Maluccio JA, Mbuya MN, Ntozini R, Tielsch JM. Plasma Concentrations of Hepcidin in Anemic Zimbabwean Infants. PLoS One. 2015 Aug 7;10(8):e0135227. doi: 10.1371/journal.pone.0135227. eCollection 2015. PMID 26252205
- [Background] Gough EK, Stephens DA, Moodie EE, Prendergast AJ, Stoltzfus RJ, Humphrey JH, Manges AR. Linear growth faltering in infants is associated with Acidaminococcus sp. and community-level changes in the gut microbiota. Microbiome. 2015 Jun 13;3:24. doi: 10.1186/s40168-015-0089-2. eCollection 2015. PMID 26106478
- [Background] Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team; Humphrey JH, Jones AD, Manges A, Mangwadu G, Maluccio JA, Mbuya MN, Moulton LH, Ntozini R, Prendergast AJ, Stoltzfus RJ, Tielsch JM. The Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial: Rationale, Design, and Methods. Clin Infect Dis. 2015 Dec 15;61 Suppl 7(Suppl 7):S685-702. doi: 10.1093/cid/civ844. PMID 26602296
- [Background] Mbuya MN, Tavengwa NV, Stoltzfus RJ, Curtis V, Pelto GH, Ntozini R, Kambarami RA, Fundira D, Malaba TR, Maunze D, Morgan P, Mangwadu G, Humphrey JH; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Design of an Intervention to Minimize Ingestion of Fecal Microbes by Young Children in Rural Zimbabwe. Clin Infect Dis. 2015 Dec 15;61 Suppl 7(Suppl 7):S703-9. doi: 10.1093/cid/civ845. PMID 26602297
- [Background] Desai A, Smith LE, Mbuya MN, Chigumira A, Fundira D, Tavengwa NV, Malaba TR, Majo FD, Humphrey JH, Stoltzfus RJ; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. The SHINE Trial Infant Feeding Intervention: Pilot Study of Effects on Maternal Learning and Infant Diet Quality in Rural Zimbabwe. Clin Infect Dis. 2015 Dec 15;61 Suppl 7(Suppl 7):S710-5. doi: 10.1093/cid/civ846. PMID 26602298
- [Background] Ntozini R, Marks SJ, Mangwadu G, Mbuya MN, Gerema G, Mutasa B, Julian TR, Schwab KJ, Humphrey JH, Zungu LI; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Using Geographic Information Systems and Spatial Analysis Methods to Assess Household Water Access and Sanitation Coverage in the SHINE Trial. Clin Infect Dis. 2015 Dec 15;61 Suppl 7(Suppl 7):S716-25. doi: 10.1093/cid/civ847. PMID 26602299
- [Background] Prendergast AJ, Humphrey JH, Mutasa K, Majo FD, Rukobo S, Govha M, Mbuya MN, Moulton LH, Stoltzfus RJ; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Assessment of Environmental Enteric Dysfunction in the SHINE Trial: Methods and Challenges. Clin Infect Dis. 2015 Dec 15;61 Suppl 7(Suppl 7):S726-32. doi: 10.1093/cid/civ848. PMID 26602300
- [Background] Mbuya MN, Jones AD, Ntozini R, Humphrey JH, Moulton LH, Stoltzfus RJ, Maluccio JA; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Theory-Driven Process Evaluation of the SHINE Trial Using a Program Impact Pathway Approach. Clin Infect Dis. 2015 Dec 15;61 Suppl 7(Suppl 7):S752-8. doi: 10.1093/cid/civ716. PMID 26602304
- [Background] Mbuya MN, Humphrey JH. Preventing environmental enteric dysfunction through improved water, sanitation and hygiene: an opportunity for stunting reduction in developing countries. Matern Child Nutr. 2016 May;12 Suppl 1(Suppl 1):106-20. doi: 10.1111/mcn.12220. Epub 2015 Nov 6. PMID 26542185
- [Background] Smith LE, Prendergast AJ, Turner PC, Humphrey JH, Stoltzfus RJ. Aflatoxin Exposure During Pregnancy, Maternal Anemia, and Adverse Birth Outcomes. Am J Trop Med Hyg. 2017 Apr;96(4):770-776. doi: 10.4269/ajtmh.16-0730. PMID 28500823
- [Derived] Piper JD, Mazhanga C, Mwapaura M, Mapako G, Mapurisa I, Mashedze T, Munyama E, Kuona M, Mashiri T, Sibanda K, Matemavi D, Tichagwa M, Nyoni S, Saidi A, Mangwende M, Mbewe G, Chidhanguro D, Mpofu E, Tome J, Mutasa B, Chasekwa B, Njovo H, Nyachowe C, Muchekeza M, Sauramba V, Gladstone MJ, Wells JC, Allen E, Moulton LH, Smuk M, Humphrey JH, Langhaug LF, Tavengwa NV, Ntozini R, Prendergast AJ. School-age growth and development following infant feeding and/or water, sanitation, and hygiene interventions in rural Zimbabwe: long-term follow-up of a cluster-randomised trial. EClinicalMedicine. 2024 Nov 22;78:102946. doi: 10.1016/j.eclinm.2024.102946. eCollection 2024 Dec. PMID 39640932
- [Derived] Piper JD, Mazhanga C, Mwapaura M, Mapako G, Mapurisa I, Mashedze T, Munyama E, Kuona M, Mashiri T, Sibanda K, Matemavi D, Tichagwa M, Nyoni S, Saidi A, Mangwende M, Chidhanguro D, Mpofu E, Tome J, Mbewe G, Mutasa B, Chasekwa B, Njovo H, Nyachowe C, Muchekeza M, Mutasa K, Sauramba V, Evans C, Gladstone MJ, Wells JC, Allen E, Smuk M, Humphrey JH, Langhaug LF, Tavengwa NV, Ntozini R, Prendergast AJ. Growth, physical, and cognitive function in children who are born HIV-free: School-age follow-up of a cluster-randomised trial in rural Zimbabwe. PLoS Med. 2024 Oct 11;21(10):e1004347. doi: 10.1371/journal.pmed.1004347. eCollection 2024 Oct. PMID 39392862
- [Derived] Evans C, Mutasa K, Rukobo S, Govha M, Mushayanembwa P, Chasekwa B, Majo FD, Tavengwa NV, Broad J, Noble C, Gough EK, Kelly P, Bourke CD, Humphrey JH, Ntozini R, Prendergast AJ. Inflammation and cytomegalovirus viremia during pregnancy drive sex-differentiated differences in mortality and immune development in HIV-exposed infants. Nat Commun. 2024 Apr 17;15(1):2909. doi: 10.1038/s41467-023-44166-2. PMID 38632279
- [Derived] Noble C, Mooney C, Makasi R, Ntozini R, Majo FD, Church JA, Tavengwa NV, Prendergast AJ, Humphrey JH; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Antenatal and delivery practices and neonatal mortality amongst women with institutional and non-institutional deliveries in rural Zimbabwe: observational data from a cluster randomized trial. BMC Pregnancy Childbirth. 2022 Dec 30;22(1):981. doi: 10.1186/s12884-022-05282-x. PMID 36585673
- [Derived] Mutasa K, Ntozini R, Mbuya MNN, Rukobo S, Govha M, Majo FD, Tavengwa N, Smith LE, Caulfield L, Swann JR, Stoltzfus RJ, Moulton LH, Humphrey JH, Gough EK, Prendergast AJ. Biomarkers of environmental enteric dysfunction are not consistently associated with linear growth velocity in rural Zimbabwean infants. Am J Clin Nutr. 2021 May 8;113(5):1185-1198. doi: 10.1093/ajcn/nqaa416. PMID 33740052
- [Derived] Ntozini R, Chandna J, Evans C, Chasekwa B, Majo FD, Kandawasvika G, Tavengwa NV, Mutasa B, Mutasa K, Moulton LH, Humphrey JH, Gladstone MJ, Prendergast AJ; SHINE Trial Team. Early child development in children who are HIV-exposed uninfected compared to children who are HIV-unexposed: observational sub-study of a cluster-randomized trial in rural Zimbabwe. J Int AIDS Soc. 2020 May;23(5):e25456. doi: 10.1002/jia2.25456. PMID 32386127
- [Derived] Chandna J, Ntozini R, Evans C, Kandawasvika G, Chasekwa B, Majo F, Mutasa K, Tavengwa N, Mutasa B, Mbuya M, Moulton LH, Humphrey JH, Prendergast A, Gladstone M. Effects of improved complementary feeding and improved water, sanitation and hygiene on early child development among HIV-exposed children: substudy of a cluster randomised trial in rural Zimbabwe. BMJ Glob Health. 2020 Jan 13;5(1):e001718. doi: 10.1136/bmjgh-2019-001718. eCollection 2020. PMID 32133164
- [Derived] Evans C, Chasekwa B, Ntozini R, Majo FD, Mutasa K, Tavengwa N, Mutasa B, Mbuya MNN, Smith LE, Stoltzfus RJ, Moulton LH, Humphrey JH, Prendergast AJ; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Mortality, Human Immunodeficiency Virus (HIV) Transmission, and Growth in Children Exposed to HIV in Rural Zimbabwe. Clin Infect Dis. 2021 Feb 16;72(4):586-594. doi: 10.1093/cid/ciaa076. PMID 31974572
- [Derived] Murenjekwa W, Makasi R, Ntozini R, Chasekwa B, Mutasa K, Moulton LH, Tielsch JM, Humphrey JH, Smith LE, Prendergast AJ, Bourke CD. Determinants of Urogenital Schistosomiasis Among Pregnant Women and its Association With Pregnancy Outcomes, Neonatal Deaths, and Child Growth. J Infect Dis. 2021 Apr 23;223(8):1433-1444. doi: 10.1093/infdis/jiz664. PMID 31832636
- [Derived] Church JA, Rogawski McQuade ET, Mutasa K, Taniuchi M, Rukobo S, Govha M, Lee B, Carmolli MP, Chasekwa B, Ntozini R, McNeal MM, Moulton LH, Kirkpatrick BD, Liu J, Houpt ER, Humphrey JH, Platts-Mills JA, Prendergast AJ. Enteropathogens and Rotavirus Vaccine Immunogenicity in a Cluster Randomized Trial of Improved Water, Sanitation and Hygiene in Rural Zimbabwe. Pediatr Infect Dis J. 2019 Dec;38(12):1242-1248. doi: 10.1097/INF.0000000000002485. PMID 31738342
- [Derived] Mbuya MNN, Matare CR, Tavengwa NV, Chasekwa B, Ntozini R, Majo FD, Chigumira A, Chasokela CMZ, Prendergast AJ, Moulton LH, Stoltzfus RJ, Humphrey JH; SHINE Trial Team. Early Initiation and Exclusivity of Breastfeeding in Rural Zimbabwe: Impact of a Breastfeeding Intervention Delivered by Village Health Workers. Curr Dev Nutr. 2019 Feb 28;3(4):nzy092. doi: 10.1093/cdn/nzy092. eCollection 2019 Apr. PMID 30937421
- [Derived] Gladstone MJ, Chandna J, Kandawasvika G, Ntozini R, Majo FD, Tavengwa NV, Mbuya MNN, Mangwadu GT, Chigumira A, Chasokela CM, Moulton LH, Stoltzfus RJ, Humphrey JH, Prendergast AJ; SHINE Trial Team. Independent and combined effects of improved water, sanitation, and hygiene (WASH) and improved complementary feeding on early neurodevelopment among children born to HIV-negative mothers in rural Zimbabwe: Substudy of a cluster-randomized trial. PLoS Med. 2019 Mar 21;16(3):e1002766. doi: 10.1371/journal.pmed.1002766. eCollection 2019 Mar. PMID 30897095
- [Derived] Church JA, Rukobo S, Govha M, Lee B, Carmolli MP, Chasekwa B, Ntozini R, Mutasa K, McNeal MM, Majo FD, Tavengwa NV, Moulton LH, Humphrey JH, Kirkpatrick BD, Prendergast AJ. The Impact of Improved Water, Sanitation, and Hygiene on Oral Rotavirus Vaccine Immunogenicity in Zimbabwean Infants: Substudy of a Cluster-randomized Trial. Clin Infect Dis. 2019 Nov 27;69(12):2074-2081. doi: 10.1093/cid/ciz140. PMID 30770931
- [Derived] Prendergast AJ, Chasekwa B, Evans C, Mutasa K, Mbuya MNN, Stoltzfus RJ, Smith LE, Majo FD, Tavengwa NV, Mutasa B, Mangwadu GT, Chasokela CM, Chigumira A, Moulton LH, Ntozini R, Humphrey JH; SHINE Trial Team. Independent and combined effects of improved water, sanitation, and hygiene, and improved complementary feeding, on stunting and anaemia among HIV-exposed children in rural Zimbabwe: a cluster-randomised controlled trial. Lancet Child Adolesc Health. 2019 Feb;3(2):77-90. doi: 10.1016/S2352-4642(18)30340-7. Epub 2018 Dec 18. PMID 30573417
- [Derived] Humphrey JH, Mbuya MNN, Ntozini R, Moulton LH, Stoltzfus RJ, Tavengwa NV, Mutasa K, Majo F, Mutasa B, Mangwadu G, Chasokela CM, Chigumira A, Chasekwa B, Smith LE, Tielsch JM, Jones AD, Manges AR, Maluccio JA, Prendergast AJ; Sanitation Hygiene Infant Nutrition Efficacy (SHINE) Trial Team. Independent and combined effects of improved water, sanitation, and hygiene, and improved complementary feeding, on child stunting and anaemia in rural Zimbabwe: a cluster-randomised trial. Lancet Glob Health. 2019 Jan;7(1):e132-e147. doi: 10.1016/S2214-109X(18)30374-7. PMID 30554749